CLINICAL TRIAL: NCT03165929
Title: Oral Flurbiprofen Spray for Mucosal Graft Harvesting at the Palatal Area: A Randomized Placebo-controlled Study
Brief Title: Oral Flurbiprofen Spray for Mucosal Graft Harvesting at the Palatal Area
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sıla Çağrı İşler, PhD, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36290600/66
Record Dates: First submitted 2017-05-21; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Surgery, Oral
Keywords: free gingival grafts; connective tissue grafts; flurbiprofen
MeSH Terms: interventions — Flurbiprofen

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- flurbiprofen-free gingival graft (Active Comparator)
  Interventions: Drug: Flurbiprofen
- placebo-free gingival graft (Placebo Comparator)
  Interventions: Drug: placebo
- flurbiprofen-connective tissue graft (Active Comparator)
  Interventions: Drug: Flurbiprofen
- placebo-connective tissue graft (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Flurbiprofen — oral flurbiprofen spray
  Arms: flurbiprofen-connective tissue graft; flurbiprofen-free gingival graft
Drug: placebo — oral placebo spray
  Arms: placebo-connective tissue graft; placebo-free gingival graft

SUMMARY:
Connective tissue graft (CTG) and free gingival graft (FGG) harvesting from the palatal area has been used frequently in the periodontal mucogingival surgery and reported to provide higher predictability and success regarding esthetic outcomes. The aim of the study was to evaluate the effects of oral flurbiprofen spray on wound healing, postoperative patient morbidity and discomfort after palatal graft harvesting.

Forty eight patients scheduled for CTG and FGG requiring periodontal plastic surgeries were selected. The patients were randomly assigned to each group, and used oral spray of flurbiprofen or placebo 3 times a day for a week. The palatal donor area was evaluated at 1 and 3 days and 1, 2, 3, 4, 6 and 8 weeks postsurgery for postoperative pain, complete epithelization, feeding habits, color match, and total number of analgesic pills taken. The Wound-Healing Index (WHI) was recorded at 2-week follow up.

DETAILED DESCRIPTION:
The palatal area, which is mostly used for connective tissue graft (SCTG) and free gingival graft (FGG) harvesting, usually provides sufficient donor tissue for periodontal plastic surgery. Surgical techniques using these procedures have been reported to present higher predictability and long term stability regarding root coverage, keratinized tissue width and soft tissue thickness increase.

Graft harvesting from the palatal area has been suggested to have some complications in the literature. Excessive hemorrhage, prolonged severe pain or discomfort, infection or necrosis of palatal tissue have been reported to occur post-operatively. To prevent these postoperative complications in the donor sites, hemostatic dressing, bioactive materials such as collagen membranes and platelet concentrates, biostimulant procedures such as low-level laser therapy and chemotherapeutic agents have been suggested. However, there is no consensus about which procedure is more efficient to reduce post-operative symptoms and to enhance early wound healing after palatal graft harvesting.

Non-steroidal anti-inflammatory drugs (NSAIDs) are the analgesic agents which widely used for the treatment of inflammation and pain management. Flurbiprofen, a chiral NSAID of the 2-arylpropionic acid class, inhibits cyclooxygenase-1 and -2 resulting in the reduced formation of prostaglandins, thromboxanes, and prostacyclin, with gastrointestinal tolerance considered better than aspirin and indomethacin, and comparable to ibuprofen and naproxen. It has been shown to possess an adequate analgesic/anti-inflammatory activity in rheumatology, gynecology, obstetrics, and oncology.

Epidemiologic studies demonstrated that systemic administration of NSAIDs commonly associated with side effects related to the gastrointestinal and renal systems. To limit the systemic exposure to oral NSAIDs and to maximize drug levels at the site of affected area, topical NSAIDs have been suggested to use. Topical flurbiprofen was reported to decrease corneal sensitivity, to effect symptomatic relief of sore throat and to reduce acute post-operative pain after oral surgical procedures in previous studies. An oral spray formulation containing 0.075 g of flurbiprofen per 30 ml spray has been developed and frequently use for the inflammatory affections of the oral cavity, pharynx and larynx.

The hypotheses for this study were that flurbiprofen spray could accelerate wound healing and reduce the patient discomfort. Therefore, the objective of the present study was to assess clinical efficacy of flurbiprofen spray on early wound healing and patient morbidity at both FGG and SCTG palatal donor sites.

ELIGIBILITY:
Inclusion Criteria:

1. age > 18 years,
2. not having any systemic disease that could compromise wound healing,
3. no periodontal surgery on the experimental sites before,
4. no smoking,
5. no pregnancy or lactation.

Exclusion Criteria:

1. hypersensitivity to flurbiprofen,
2. history of allergy to NSAIDs,
3. having coagulation disorders,
4. presence of gagging reflex.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
complete epithelization | 2 months postoperatively
  the time needed to obtain complete epithelization of the palatal wounds

SECONDARY OUTCOMES:
patients' discomfort | 2 months postoperatively
  Visual Analogue Scale (VAS)
postoperative swelling | 2 months postoperatively
  Visual Analogue Scale (VAS)
changes in patients' feeding habits | 2 months postoperatively
  Visual Analogue Scale (VAS)
burning sensation | 2 months postoperatively
  Visual Analogue Scale (VAS)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Isler SC, Eraydin N, Akkale H, Ozdemir B. Oral flurbiprofen spray for mucosal graft harvesting at the palatal area: A randomized placebo-controlled study. J Periodontol. 2018 Oct;89(10):1174-1183. doi: 10.1002/JPER.17-0381. Epub 2018 Aug 29. PMID 30007054